CLINICAL TRIAL: NCT03293914
Title: Addressing Uncontrolled Diabetes in Primary Care: A Lifestyle Redesign Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Los Angeles County Department of Health Services (DHS) (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Beth Pyatak, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC CTSI Grant #UL1TR001855; UL1TR001855 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-09-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: This is an implementation trial being conducted in a real-world clinical setting in which masking is not appropriate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be invited to enroll in an occupational therapy (OT) lifestyle redesign intervention focused on diabetes management. The intervention includes approximately 8 one-hour OT sessions over 4 months.
  Interventions: Behavioral: Lifestyle Redesign
- Usual Care Control (No Intervention): Participants will not be contacted; outcome data will be extracted from medical records.

INTERVENTIONS:
Behavioral: Lifestyle Redesign — Individualized lifestyle intervention incorporating the following topics: Diabetes knowledge; access to healthcare; communication with healthcare providers; incorporation of diabetes self-care tasks within daily habits and routines; social support; and emotional well-being. Participants receive approximately 8 hours of intervention by a licensed occupational therapist with training in diabetes education, motivational interviewing and the intervention protocol.
  Other Names: Resilient, Empowered, Active Living with Diabetes (REAL)
  Arms: Intervention

SUMMARY:
This study is examining the feasibility of implementing an occupational therapy intervention addressing diabetes management in a primary care clinic within the Los Angeles County Department of Health Services (LAC-DHS), as well as the impact of this intervention approach on clinical outcomes, efficiency and patient-centeredness of care. This implementation science study is evaluating two emerging trends in healthcare delivery: (1) the integration of nontraditional providers into primary care medical home (PCMH) settings to facilitate the delivery of high-quality, comprehensive primary care while reducing the burden on physicians; and (2) the potential value of using occupational therapists to address chronic disease management in this setting

ELIGIBILITY:
Inclusion Criteria:

* Current patient at Los Angeles County-USC Medical Center Adult West Primary Care clinic
* Diagnosed diabetes (type 1 or type 2) documented in EMR
* Most recent HbA1c level >9.0% OR has not had an HbA1c measurement within past 12 months
* Per provider judgment, would be willing to make lifestyle changes related to diabetes self-care

Exclusion Criteria:

* Active, untreated substance use or behavioral health disorder which interferes with participation in major life activities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in the daily rate of change of Glycated hemoglobin (HbA1C) during the year prior to baseline, compared to the period from baseline to post-intervention | all measures taken from one year prior to baseline, to immediately post-intervention (an average of 4 months)
  Measure of average blood glucose concentration over approximately the previous 12 weeks. HbA1C is measured periodically, as prescribed by study-independent provider.

SECONDARY OUTCOMES:
Change from baseline in Audit of Diabetes-Dependent Quality of Life (ADD-QoL) at post-intervention | Baseline, an average of 4 months
  19-item survey measure assessing impact of diabetes on social, physical, and emotional functioning.
Difference in the daily rate of change of Patient Health Questionnaire-9 (PHQ-9) during the year prior to baseline, compared to the period from baseline to post-intervention | all measures taken from one year prior to baseline, to immediately post-intervention (an average of 4 months)
  9-item survey measure assessing severity of depressive symptoms. PHQ-9 is measured at each study-independent clinic visit for patients who screen positive on the PHQ-2 (score >2).
Change from baseline in Summary of Diabetes Self-Care Activities (SDSCA) at post-intervention | Baseline, an average of 4 months
  14 items assessing diet, physical activity, medication adherence and other self-care behaviors relevant to diabetes.
Change from baseline in Medication adherence scale at post-intervention | Baseline, an average of 4 months
  3-item self-report medication adherence scale designed by Ira B. Wilson, Yoojin Lee, Joanne Michaud, Floyd J. FowlerJr., and William H. Rogers
Change from baseline in Appraisal of Diabetes Scale at post-intervention | Baseline, an average of 4 months
  7-item self-report scale assessing the individual's appraisal of his or her diabetes
Change from baseline RAND 20-Item Short Form Survey (SF-20) at post-intervention | Baseline, an average of 4 months
  The SF-20 is a 20-item set of generic, coherent, and easily administered quality-of-life measures.
Acceptability | Months 11-12
  Both formative and summative data will be gathered throughout the study to assess acceptability, defined herein as the perception of the intervention as agreeable/satisfactory. Acceptability will be assessed through interviews.
Appropriateness | Months 0-2, 3-10, and 11-12
  Both formative and summative data will be gathered throughout the study to assess appropriateness, defined herein as the perceived relevance or compatibility of the intervention in the practice setting. Appropriateness will be assessed through interviews.
Feasibility | Months 0-2, and 11-12
  Both formative and summative data will be gathered throughout the study to assess feasibility, defined herein as the extent to which the intervention can be successfully used in a practice setting. Feasibility will be assessed through surveys.
Fidelity | Months 0-2, 3-10, and 11-12
  Both formative and summative data will be gathered throughout the study to assess fidelity, defined herein as the extent to which the intervention is implemented as intended. Fidelity will be assessed through score on fidelity checklist.
Efficiency | Months 0-2 and 11-12
  Both formative and summative data will be gathered throughout the study to assess efficiency, defined herein as the degree to which providers work to the "top of license". Efficiency will be assessed through interviews.
Timeliness | Months 11-12
  Both formative and summative data will be gathered throughout the study to assess timeliness, defined herein as the availability of appointments when needed. Timeliness will be assessed through staff documentation records.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pyatak, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Primary Care Adult West Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No